# Relationship and sexual satisfaction of stoma patients 18.04.2022

NCT ID: konstanz\_001

Study protocol

18.04.2022 

# Relationship and sexual satisfaction of stoma patients – study protocol

# 18.04.2022

# **Version 2**

Head of study: Dr. med. Silvan Hämmerli

deputy: Prof. Dr. med. Jörg Glatzle

# **Table of contents**

| 1. | Background | 3 |
|----|----------------------------|---|
| 2. | Aim | 3 |
| 3. | Participants | 3 |
| 4. | Methods | 3 |
| 5. | Statistics | 3 |
| 6. | Protection of data privacy | 3 |
| 7. | Risks | 3 |
| 8. | References | 3 |

18.04.2022 

### 1 Background

Sexual dysfunctions are common after stoma operations with rectal cancer. <sup>1</sup> Sexual dysfunctions after rectum operations are a known complication. <sup>2</sup> Pateints with stoma have a significantly lower self-esteem compared to helathy people. <sup>3</sup> There is no research regarding the connection of a stoma and sexual satisfaction to the best of our knowledge. To advise patients before such an operation it is necessary to investigate such a connection.

#### 2 Aim

- Sexual satisfaction of participants with stoma
- Relationship satisfaction of participants with stoma
- Comparing colostomy and ileostomy
- Sesensitize people treating patients with stoma

#### 3 Patients

Patients with stoma or after having had a stoma are asked to fill out an online questionnaire regarding sexual and relationship satisfaction.

Minimum age: 18 years

No sexual dysfunctions. No disease influencing sexual functioning

#### 4 Methods

Anonymous Questionnaire. Retrospective data analysis.

#### 5 Statistics

Empiric data analysis of answers and comparing answers to literature.

#### 6 Protection of data privacy

Questionnaire is anonymous. Data is only avaliable with password. Only head of study and deputy have access to data.

#### 7 Risks

The study is an anonymous questionnaire. The data is analysed retrospectively. So there are no risks for participants.

#### 8 References

- 1. Sutsunbuloglu, E., & Vural, F. (2018). Evaluation of sexual satisfaction and function in patients following stoma surgery: A descriptive study. *Sexuality and Disability*, *36*(4), 349-361.
- 2. Hendren, S. K., O'Connor, B. I., Liu, M., Asano, T., Cohen, Z., Swallow, C. J., ... & McLeod, R. S. (2005). Prevalence of male and female sexual dysfunction is high following surgery for rectal cancer. *Annals of surgery*, *242*(2), 212.

18.04.2022 

3. Gozuyesil, E., Taylan, S., Manav, A. I., & Akil, Y. (2017). The evaluation of self-esteem and sexual satisfaction of patients with bowel stoma in Turkey. *Sexuality and Disability*, *35*(2), 157-169.

18.04.2022 